CLINICAL TRIAL: NCT03796130
Title: Does Myomectomy for Intramural Fibroid Improve ART Outcome? A Randomized Controlled Trial
Brief Title: Does Myomectomy for Intramural Fibroid Improve ART Outcome?
Acronym: MIFART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Collaborators: Alexandria University (Other); Zagazig University (Other Government); Sohag University (Other); Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gibreel, Assistant professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H0008
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-11

CONDITIONS: Fibroid Uterus
MeSH Terms: conditions — Leiomyoma | interventions — Uterine Myomectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (A)Myomectomy (Experimental): This study will include women who have intramural myomas ranging from 3-5 cm
  The participants will be randomlyallocated intotwo groups.
  In group (A): myomectomy will be performed before ART
  In group 1, ART will be performed 3 months after myomectomy if the uterine cavity is not opened and 6 months after myomectomy upon inadvertent opening of the uterine cavity during surgery
  Interventions: Procedure: Myomectomy
- (B) No myomectomy (No Intervention): This study will include women who have intramural myomas ranging from 3-5 cm
  The participants will be randomly allocated into two groups.
  In group (B):women will have their trial of ART without myomectomy

INTERVENTIONS:
Procedure: Myomectomy — This study will include women who have intramural myomas ranging from 3-5 cm
  The participants will be randomly allocated into two groups.
  In group (1): myomectomy will be performed before ART
  In group (2):women will have their trial of ART without myomectomy
  In group A, ART will be performed 3 months after myomectomy if the uterine cavity is not opened and 6 months after myomectomy upon inadvertent opening of the uterine cavity during surgery
  Arms: (A)Myomectomy

SUMMARY:
Intamural fibroids (myoma) do exist in some infertile women undergoing IVF treatment. There is controversy whether myomectomy before IVF treatment could improve IVF outcome. This trial will examine whether myomectomy in those patients could improve the results.

DETAILED DESCRIPTION:
This study will include women who have intramural myoma ranging from 3-5 cm

The participants will be randomly allocated into two groups.

In group (1): myomectomy will be performed before ART

In group (2):women will have their trial of ART without myomectomy

In group A, ART will be performed 3 months after myomectomy if the uterine cavity is not opened and 6 months after myomectomy upon inadvertent opening of the uterine cavity during surgery

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* Women with intramural fibroid without any cavity involvement
* Age ˂ 35 years
* I onCSI or IVF cycles
* normal uterine cavity

Exclusion Criteria:

* Exclusion criteria:
* low ovarian reserve (AFC < 7 and or AMH < 1.1 ng/ml)
* Endometrioma
* Untreated hydrosalpinx
* Non obstructive azoospermia
* Any other cavitary lesions (Asherman syndrome, Mullerian anomalies)
* recurrent implantation failure

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 80 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be ongoing pregnancy rate | 3 months after embryo transfer
  Pregnancy continued after 12 week gestation per randomised women

SECONDARY OUTCOMES:
-Implantation rate | 15 days after embryo transfer
-clinical pregnancy rate | 5 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gibreel, MD, Principal Investigator — Mansoura University; Mohamed S Abdelhafez, MD, Study Director — Mansoura University; Salah Rasheed, MD, Study Director — Sohag University; Ahmed Nasr, MD, Study Director — Assiut Universit; Hisham A Saleh, MD, Study Director — Alexandria University; Hassan El Maghraby, MD, Study Director — Alexandria University; Eman El Gindy, MD, Study Chair — Zagazig University; Hoda Sibai, MD, Study Director — Zagazig University; Hamed Yossef, MD, Study Chair — Mansoura University
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes